CLINICAL TRIAL: NCT04845776
Title: Vitamin/Mineral Supplement for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Southwest College of Naturopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00013694
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: All study participants with ASD will receive the vitamin/mineral supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This group receives the vitamin/mineral supplement, ANRC Essentials Plus, for 3 months
  Interventions: Dietary Supplement: ANRC Essentials Plus

INTERVENTIONS:
Dietary Supplement: ANRC Essentials Plus — a vitamin/mineral supplement designed for children and adults with autism

SUMMARY:
This is an open-label 3 month clinical trial of a vitamin/mineral supplement designed for children with autism.

DETAILED DESCRIPTION:
This is an open-label 3 month clinical trial of a vitamin/mineral supplement designed for children with autism. There will be pre/post assessments of autism symptoms,GI symptoms, and laboratory tests. Typically-developing children will be assessed at baseline only (no treatments) for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Child age 3-17 years (up until 18th birthday)
2. Previous diagnosis of ASD by a psychiatrist, psychologist, or developmental pediatrician
3. Verification of diagnosis by ASU staff using the Autism Diagnostic Interview-Revised.
4. No changes in any medical, nutritional, dietary, behavior, or other treatment in the last three months, and a willingness to avoid any changes during the study
5. Participant is able to wear a mask during the short visit for the blood draw.

Exclusion Criteria:

1. Parent/guardian is unable to read or speak English fluently.
2. Use of a vitamin/mineral supplement in the past 3 months
3. Previous adverse reaction to a vitamin/mineral supplement
4. Unstable, poor health; seizure disorder that is not responsive to treatment or not on stable management or complex type; or other health conditions that would significantly increase their risk of adverse effects (per physician clinical judgement)
5. Use of any medication which has a contra-indication for one of the ingredients in the vitamin/mineral supplement
6. A major single-gene disorder such as Fragile X, Down's Syndrome.
7. Major brain malformation
8. Tube feeding
9. Current participation in other clinical trials
10. Females who are pregnant or who are sexually active without effective birth control.
11. Clinically significant abnormalities at baseline on two blood safety tests: Comprehensive Metabolic Panel and Complete Blood Count with Differential.
12. Psychotropic medication use which can affect neurotransmitter levels/function - Current or within past 2 months

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Parent Global Impressions of Autism | assessed at the 3 months (end of treatment)
  a 20-item questionnaire with a Likert scale assessing changes in symptoms

CONTACTS AND LOCATIONS:
Overall Officials: James B Adams, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website for our research group — http://autism.asu.edu